CLINICAL TRIAL: NCT02103140
Title: An Exercise Randomized Controlled Trial Targeting African-American Women With Metabolic Syndrome and High Risk for Breast Cancer
Brief Title: An Exercise RCT Targeting African-American Women With Metabolic Syndrome and High Risk for Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2012-012 Georgetown Lombardi
Record Dates: First submitted 2014-04-01; First posted 2014-04-03 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: Breast Cancer; Obesity; African American female; exergaming
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Facility-Based Exercise Intervention (Experimental): Supervised Facility-Based Exercise Intervention Arm The participants randomized to the exercise group will be required to meet and maintain a goal of 150 min/wk of moderate intensity exercise for 6 months. This intervention will use heart rate and rating of perceived exertion (RPE) to define moderate intensity. Participants will exercise for the prescribed duration at a heart rate in the range of 45-65% of their maximal oxygen consumption (VO2 max), as determined during baseline testing, and with an RPE in the range of 11-14 on the 20-point scale. The exercise will primarily utilize treadmills and exercise bikes.
  Interventions: Behavioral: Facility-based Exercise
- Control (No Intervention): After baseline testing, the control group will be asked to maintain their current daily activities and exercise habits for the duration of the study (6 months). The control group will have measurements at the same time periods as the participants in the intervention arm through the completion of the study. Participants will be seen for follow-up at 3 and 6 months (study completion). The participants in the control group will receive the same incentives as those in the intervention arms (gift cards). Since the women in the control group are obese, with components of metabolic syndrome, and at relatively high risk for breast cancer, we are providing healthy lifestyle information to the group, via text messages.
- Home-Based Exercise Intervention (Experimental): Home-Based Exercise Intervention Group The participants randomized to this intervention arm will be required to meet and maintain a goal of 150 min/wk of moderate intensity exercise for 6 months, the same as the supervised intervention group. Their exercise goal will be to achieve a total of 10,000 steps per day, as measured by pedometers. Participants will be required to have a cell phone with text messaging capabilities.
  Interventions: Behavioral: Home-based Exercise

INTERVENTIONS:
Behavioral: Facility-based Exercise — Supervised Facility-Based Exercise Intervention Arm The participants randomized to the exercise group will be required to meet and maintain a goal of 150 min/wk of moderate intensity exercise for 6 months. This intervention will use heart rate and rating of perceived exertion (RPE) to define moderate intensity. Participants will exercise for the prescribed duration at a heart rate in the range of 45-65% of their maximal oxygen consumption (VO2 max), as determined during baseline testing, and with an RPE in the range of 11-14 on the 20-point scale. The exercise will primarily utilize treadmills and exercise bikes.
  Arms: Facility-Based Exercise Intervention
Behavioral: Home-based Exercise — Home-Based Exercise Intervention Group The participants randomized to this intervention arm will be required to meet and maintain a goal of 150 min/wk of moderate intensity exercise for 6 months, the same as the supervised intervention group. Their exercise goal will be to achieve a total of 10,000 steps per day, as measured by pedometers. Participants will be required to have a cell phone with text messaging capabilities.
  Arms: Home-Based Exercise Intervention

SUMMARY:
Among African-American women, in whom metabolic syndrome (MetS) is very prevalent and breast cancer mortality rates are high, it is hypothesized that intervening on MetS to improve the MetS profile may prove to be a means to reduce breast cancer risk. Specific recommendations for breast cancer prevention are now focused on maintaining a healthy weight via increased physical activity levels, and losing weight if overweight or obese.

This pilot project compares two exercise interventions: a supervised facility-based and a home-based exercise intervention to a control group in African-American women with metabolic syndrome who are at high risk for breast cancer. This study is a 6-month three-arm RCT to assess the impact of the exercise interventions on biomarkers related to obesity, insulin-related pathways, inflammation, hormones, and micro-RNAs.

The specific aim of the proposed study is to compare the impact of a supervised facility-based and a home-based exercise intervention on obesity, metabolic syndrome and known breast cancer biomarkers in postmenopausal African-American women with metabolic syndrome who are at increased risk of breast cancer.

DETAILED DESCRIPTION:
1. To assess the impact of exercise on biomarkers related to obesity, insulin-related pathways, inflammation, hormones, and microRNAs.
2. The primary aim of this study is to compare the effect of 2 types of exercise interventions (supervised and self-directed compared to control) on biological parameters related to breast cancer development. It is important to understand if participants in this study respond better to an exercise program they are able to engage in on their own (self-directed) or if participating in an exercise program under supervision is preferred. A study by Pinto utilized a home-based exercise program among breast cancer survivors and commented that the home-based program has several advantages including 1) mitigating transportation and scheduling difficulties, and 2) is less expensive than supervised programs. Another study compared the effect of a supervised exercise program to a self-directed exercise group and a control group on physical functioning and health-related quality of life among breast cancer survivors and found that participants in the self-directed exercise group improved their physical functioning to a somewhat greater degree than the supervised group. The authors proposed that one reason for this result could be attributed to the fact that the self-directed program included many features thought to comprise effective home training including the following: baseline fitness evaluations, written guidelines for home exercise, education about pulse checking/heart rate guidelines, daily activity logs and bi-weekly telephone calls by the exercise specialist. In the current study, we plan to employ features similar to the self-directed exercise program in an effort to determine if the self-directed group improves to a greater extent than the control group and better or comparable to the supervised group. An added feature of the current study is that we will administer a participant satisfaction questionnaire to assess each participant's experience in their respective groups. This information will, in part, help us to plan future studies. All participants will complete a baseline assessment prior to randomization, as indicated in Table 1 in the attached grant proposal; follow-up measures will also be conducted as indicated in that table. Participants will be required to provide a medical clearance from their health care provider or a nurse practitioner.
3. * Rationale and justification for study (i.e. historical background, investigator's personal experience, pertinent medical literature, etc.): In the United States, breast cancer is the most commonly diagnosed cancer in women, other than non-melanoma skin cancer, and is the second most common cause of cancer deaths among women. Several risk factors have been identified that increase breast cancer risk, some of which are non-modifiable (e.g., age, family history, and race) and some of which are modifiable (e.g., physical activity, body weight, dietary habits, and alcohol intake). Breast cancer rates, which are increasing worldwide, parallel the increases in lifestyle diseases including Type 2 diabetes, obesity, and metabolic syndrome (MetS). MetS represents a cluster of risk factors associated with increased risk of cardiovascular diseases, and includes several components individually related to breast cancer etiology, i.e., central obesity, hypertension, hyperglycemia, and low high-density lipoprotein cholesterol. However, recent studies have suggested that MetS is underdiagnosed in African-American women because they are less likely to have decreased HDL or increased triglycerides as compared to women of other races/ethnicities. Breast cancer is hormone related and thus, the effects of established risk factors for the disease, including obesity, differ before to after menopause. Among African-American women, in whom MetS is very prevalent and breast cancer mortality rates are high, it is hypothesized that intervening on MetS to improve the MetS profile may prove to be a means to reduce breast cancer risk. The American Cancer Society (ACS) and the International Agency for Research on Cancer of the World Health Organization now both recommend regular physical activity as a strategy for women to reduce their risk of developing breast cancer. Specific recommendations for breast cancer prevention, which initially emphasized diet, are now focused on maintaining a healthy weight throughout life by balancing caloric intake while increasing caloric expenditure via increased physical activity levels, and losing weight if overweight or obese.

Obesity itself is a major public health problem and is associated with increased postmenopausal breast cancer incidence and mortality. Our proposed pilot project compares two exercise interventions: a supervised facility-based and a home-based exercise intervention to a control group in African-American women with metabolic syndrome who are at high risk for breast cancer (based on the CARE model).This study is a 6-month three-arm RCT to assess the impact of the exercise interventions on biomarkers related to obesity, insulin-related pathways, inflammation, and hormones. The specific aim of the proposed study is to compare the impact of a supervised facility-based and a home-based exercise intervention on obesity, metabolic syndrome and known breast cancer biomarkers in postmenopausal African-American women with metabolic syndrome who are at increased risk of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants should be female, African-American postmenopausal women between the ages of 45 and 65 with waist circumference greater than 35 inches (88 cm), 5-year invasive breast cancer risk is greater than 1.40% using the CARE model, and have at least one of the following:
* elevated fasting glucose is greater than or equal to 100 mg/dL
* elevated blood pressure is greater than or equal to 130/85 mm/Hg. In addition, they should also have a cell phone with texting capabilities, read and speak English, reside in close proximity to, or can access the Navy Yard stop on the green line, can provide meaningful consent, and medical clearance from a physician or nurse practitioner.

Exclusion Criteria:

* -physical limitations that prevent participant from exercising
* premenopausal
* pregnant or planning to become pregnant within the next year
* history of cancer (except for non-melanoma skin cancer)
* have diabetes
* use anti-diabetic medication (including insulin)
* are currently enrolled in a physical activity and/or dietary clinical trial
* are on a weight loss program
* cannot commit to the intervention schedule

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2023-09 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Waist circumference | 6 months
  Reduction in waist circumference
Body Mass Index | 6 months
  Reduction in body mass index
Biomarkers of breast cancer risk - biomarkers of inflammation | 6 months
  Serum IL-6, TNF-alpha, High sensitivity CRP
Biomarkers of breast cancer risk - biomarkers of insulin pathway | 6 months
  Fasting glucose, seruminsulin, IGF-1, IGFBP-3
Biomarkers of breast cancer risk - adipokines | 6 months
  Serum leptin and adiponectin
Metabolic syndrome | 6 months
  Greater improvements in metabolic syndrome and metabolic syndrome components

SECONDARY OUTCOMES:
Cardiorespiratory fitness | 6 months
  VO2Max using the Bruce treadmill protocol
Body composition | 6 months
  Measured using DEXA scan: fat mass, lean mass
Health-related Quality of Life | 6 months
  Measured using the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown Lombardi Office of Minority Health community site, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Adams-Campbell LL, Taylor T, Hicks J, Lu J, Dash C. The Effect of a 6-Month Exercise Intervention Trial on Allostatic Load in Black Women at Increased Risk for Breast Cancer: the FIERCE Study. J Racial Ethn Health Disparities. 2022 Oct;9(5):2063-2069. doi: 10.1007/s40615-021-01145-x. Epub 2021 Sep 27. PMID 34580826
- [Derived] Dash C, Makambi K, Wallington SF, Sheppard V, Taylor TR, Hicks JS, Adams-Campbell LL. An exercise trial targeting African-American women with metabolic syndrome and at high risk for breast cancer: Rationale, design, and methods. Contemp Clin Trials. 2015 Jul;43:33-8. doi: 10.1016/j.cct.2015.04.015. Epub 2015 May 8. PMID 25962889